CLINICAL TRIAL: NCT07374237
Title: Evaluation of Interoception, Fatigue, and Upper and Lower Extremity Functional Capacity in Multiple Sclerosis Patients With Good and Poor Sleep Quality
Status: Recruiting | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Özge Çoban, Assistant Professor, Gulhane School of Medicine
Other Study IDs: 08/1454
Record Dates: First submitted 2026-01-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; interoception; fatigue; functional capacity; sleep quality
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 51 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis Patients with Poor Sleep Quality: Participants with a Pittsburgh Sleep Quality Index (PSQI) total score of 5 or higher, indicating poor sleep quality.
- Multiple Sclerosis Patients with Poor Good Quality: Good sleep quality group: Participants with a Pittsburgh Sleep Quality Index (PSQI) total score below 5, indicating good sleep quality.

SUMMARY:
Multiple sclerosis (MS) is a chronic disease of the central nervous system associated with a wide range of motor and non-motor symptoms. Sleep disturbances, fatigue, altered interoceptive perception, and impairments in upper and lower extremity functional capacity are commonly observed in individuals with MS. Decreased sleep quality may exacerbate fatigue and negatively affect daily activities and independence. Therefore, examining the relationships between sleep quality, interoception, fatigue, and extremity functional capacity is essential for effective disease management and the preservation of quality of life in individuals with MS.

The aim of this study is to compare interoception, fatigue, and upper and lower extremity functional capacity between individuals with MS who have good and poor sleep quality and to evaluate the relationships among these variables. By comparing MS patients based on sleep quality, this study seeks to clarify the impact of sleep quality on interoceptive processes, fatigue levels, and functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple sclerosis by a specialist physician
* Aged between 18 and 65 years
* No MS relapse within the last 3 months
* Expanded Disability Status Scale (EDSS) score between 1.0 and 5.0
* Ability to stand independently for at least 60 seconds without the use of any assistive device
* No additional neurological disorder or circulatory/visual impairment that may affect balance
* Cognitive function score >24 on the Mini-Mental State Examination (MMSE)
* Provided written informed consent after receiving detailed information about the study

Exclusion Criteria:

* Use of corticosteroids within the last 4 weeks
* Pregnancy
* Presence of spinal deformities, disc herniation, or other spinal pathologies
* Presence of orthopedic conditions affecting the hip, knee, or ankle
* History of surgery involving the spine, hip, knee, or ankle
* Change in medication within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals diagnosed with multiple sclerosis (MS) by a specialist physician. Eligible participants are adults aged 18-65 years, with an Expanded Disability Status Scale (EDSS) score between 1.0 and 5.0, who have not experienced an MS relapse within the past three months. Participants must be able to stand independently for at least 60 seconds without assistive devices and have sufficient cognitive function, defined as a Mini-Mental State Examination score greater than 24. Exclusion criteria include other neurological, visual, or circulatory conditions affecting balance, recent corticosteroid use, pregnancy, significant orthopedic or spinal disorders, and recent medication changes. Written informed consent is obtained from all participants prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index Total Score | From November 1, 2025 to June 1, 2026
  Sleep quality refers to the subjective evaluation of sleep characteristics, including sleep duration, latency, efficiency, disturbances, and daytime dysfunction, and was assessed using the Pittsburgh Sleep Quality Index (PSQI). Total scores range from 0 to 21, with higher scores indicating poorer sleep quality. A cut-off score of 5 was applied; scores greater than 5 indicate poor sleep quality, whereas scores less than 5 indicate good sleep quality.
Interoceptive Accuracy Score | From November 1, 2025 to June 1, 2026
  Interoceptive accuracy refers to the ability to accurately perceive internal bodily signals and was assessed using the Heartbeat Counting Task. During the task, participants were instructed to silently count their own heartbeats without manually checking their pulse during predefined time intervals. Simultaneously, actual heartbeats were recorded using a physiological recording device. Interoceptive accuracy was calculated by comparing the number of counted heartbeats with the recorded heartbeats. Scores range from 0 to 1, with higher scores indicating better interoceptive accuracy.
Fatigue Severity Scale Mean Score | From November 1, 2025 to June 1, 2026
  Fatigue severity refers to the perceived intensity and impact of fatigue on daily functioning and was assessed using the Fatigue Severity Scale (FSS). The FSS is a self-report questionnaire consisting of 9 items, each rated on a 7-point Likert scale. The mean score was calculated by averaging the item scores and ranges from 1 to 7, with higher scores indicating greater fatigue severity.
Multiple Sclerosis Functional Composite (MSFC) Composite Score | From November 1, 2025 to June 1, 2026
  Functional capacity refers to the ability to perform motor and cognitive tasks related to daily functioning and was assessed using the Multiple Sclerosis Functional Composite (MSFC) in patients with multiple sclerosis. The MSFC is a composite measure consisting of lower extremity function assessed by the Timed 25-Foot Walk, upper extremity function assessed by the 9-Hole Peg Test, and cognitive processing speed assessed by the Paced Auditory Serial Addition Test. Scores from each component were standardized and combined to generate a composite MSFC score, with higher scores indicating better functional capacity.
Interoceptive Awareness Scores | From November 1, 2025 to June 1, 2026
  Interoceptive awareness refers to the conscious perception and appraisal of internal bodily sensations and was assessed using the Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) questionnaire. The MAIA-2 is a self-report measure consisting of 32 items assessing multiple dimensions of interoceptive awareness. Total scores range from 0 to 160, with higher scores indicating better interoceptive awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided